CLINICAL TRIAL: NCT03893292
Title: A Pilot Study on the Utility of Cooled Radiofrequency Ablation in Patients Prior to Total Knee Arthroplasty
Brief Title: Preop Cooled Radiofrequency Ablation for Total Knee Replacement
Status: Withdrawn | Type: Observational
Why Stopped: Lack of participants
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1149
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Pain; Knee Osteoarthritis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Preoperative cooled radiofrequency ablation: Patients who undergo cooled radiofrequency ablation within 4-8 weeks of their scheduled total knee replacement.
  Interventions: Procedure: Total knee replacement; Device: COOLIEF

INTERVENTIONS:
Procedure: Total knee replacement — Patients will undergo total knee replacement surgery.
Device: COOLIEF — The superior lateral genicular nerve, superior medial genicular nerve, and inferior medial geniculate nerve will be ablated.

SUMMARY:
Total knee replacement surgery is commonly performed for patients suffering from severe knee osteoarthritis. However, 20% of patients continue to experience pain after surgery. There is currently no standardized pain management protocol for pain after total knee replacement. Cooled radiofrequency ablation has been used successfully to alleviate spin-related pain and has recently been approved by the FDA to treat chronic knee arthritic pain. This pilot study aims to collect preliminary data on the use of cooled radiofrequency ablation in patients undergoing total knee replacement.

DETAILED DESCRIPTION:
The number of patients who undergo total knee replacement is rising significantly. However, many of these patients are dissatisfied with the results, because they continue to experience pain postoperatively. This pain can be debilitating and can also be associated with decreased quality of life. Given the increasing number of patients undergoing total knee replacement and a dissatisfaction rate of 8-44%, improvements must be made in pain management protocols to help decrease pain in the immediate postoperative period following total knee replacement. Cooled radiofrequency ablation is a procedure that uses water-cooled technology to denervate the sensory nerves. It is widely used in the spine and is increasingly being used in the knee to treat osteoarthritis. Existing studies have shown that it can significantly reduce pain in patients with chronic osteoarthritis. In terms of its potential benefit as a preoperative measure to minimize postoperative pain, the literature is sparse. Results from this study will be used to generate hypotheses and power for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total knee replacement for osteoarthritis
* Pain >6 (on a scale of 0-10)
* Body mass index: 21-35 kg/m2

Exclusion Criteria:

* Age <65 years
* Patients who are wheelchair bound
* History of inflammatory arthritis or rheumatic disease
* Body mass index <21 or >35 kg/m2
* Chronic opioid use
* Pregnant women
* Non-English speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing unilateral primary total knee replacement for the treatment of knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Pain | Up to 1 year post-total knee replacement
  Pain will be assessing on a 0-10 scale, where 0=no pain and 10=most pain.

SECONDARY OUTCOMES:
Knee Disability | Up to 1 year post-total knee replacement
  Knee disability will be assessed using the Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR). The score ranges from 0-100, where 0=total knee disability and 10=perfect health.
Function assessed using the PROMIS-physical function computer adaptive test | Up to 1 year post-total knee replacement
  Function will be assessed using the PROMIS-physical function computer adaptive test. A higher score indicates higher function.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kirschner, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No